CLINICAL TRIAL: NCT03218332
Title: Post-Concussion Syndrome in Professional Athletes: A Multidisciplinary Study
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Weston A. Price Foundation (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Marion and Gerald Soloway Professorship in Brain Injury and Concussion Research,Assistant Professor, University Health Network, Toronto
Other Study IDs: 11-0088-B
Record Dates: First submitted 2017-05-01; First posted 2017-07-14 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Traumatic Encephalopathy
MeSH Terms: conditions — Chronic Traumatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid (CSF) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Former concussed pro-athletes: Biomarkers for detecting possible CTE invivo in former pro-athletes with multiple concussions: Imaging/blood/cerebrospinal fluid (CSF)/Positron emission tomography (PET-)tau/magnetic resonance imaging (MRI)/neuropsychological assessment.
  Interventions: Diagnostic Test: Biomarkers for detecting possible CTE invivo
- Healthy controls: Active Comparator
  Interventions: Diagnostic Test: Biomarkers for detecting possible CTE invivo

INTERVENTIONS:
Diagnostic Test: Biomarkers for detecting possible CTE invivo — Detection biomarkers for possible CTE: Imaging/blood/CSF/PET-tau/MRI/europsychological assessment

SUMMARY:
to examine the relationship between repeated concussions and late decline of brain function. In addition, all participants agreeing to participate in the study will be asked to will their brains to The Krembil Neuroscience Centre Concussion Project at the Toronto Western Hospital with the consent and full knowledge of their families and doctors. However, it is possible to participate in the research without agreeing to a brain donation.

The Project Team is specifically attempting a clinical-MRI-brain tissue research analysis to determine the exact mechanism of the damage to brain tissue following repeated concussions. This condition is known as chronic traumatic encephalopathy (CTE), and shows an abnormal protein in the brain called tau-protein.

DETAILED DESCRIPTION:
We hypothesize that repeated concussions in retired professional athletes will be associated with abnormalities in neurological, neuropsychological, biofluids and neuroimaging assessments. The primary objectives of the study are:

1. To determine the effects of repeated concussions on neurological, neuropsychological and psychosocial functioning.
2. To determine the relationship between repeated concussions and neuroanatomical abnormalities in brain gray and white matter subserving cognitive and motor functions using structural MRI assessment.
3. To determine the relationship between repeated concussions and changes in the cerebrospinal fluid composition.
4. To (i) establish the infrastructure to conduct ongoing pathological examination of donated brains.
5. In order to investigate whether the effects of repeated concussions on brain function and brain structure are progressive and related to the condition known as Chronic Traumatic Encephalopathy, prospective, longitudinal, follow-up data will be collected

ELIGIBILITY:
Inclusion Criteria:

fluent in English, and a history of multiple concussions , low exposures , or no concussions (Control group ). Determination of concussion exposure will be determined as follows: Previous concussion will be based on the player's recall of injury and defined as "an injury resulting from a blow to the head that caused an alteration in mental status and one or more of the following symptoms: headache, nausea, vomiting, dizziness/balance problems, fatigue, trouble sleeping, drowsiness, sensitivity to light or noise, blurred vision, difficulty remembering, and difficulty concentrating.

Exclusion Criteria:

Neurological disorders prior to concussions (e.g.: seizure disorder); systemic illnesses known to affect the brain (e.g., diabetes and lupus); a history of psychotic disorder; known developmental disorders (e.g., attention deficit disorder, dyslexia); history of migraines; and, active engagement in litigation.

Ages: 25 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retired professional athletes with history or multiple concussions and healthy control group without any history of concussion
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-07-04 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for possible CTE | several visits every two years up to 10 years
  Neuropsychological/MRI/genetics/CSF/PET-tau/oculomotor

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carmela Tartaglia, M.D, Principal Investigator — Toronto Western Hopsital,UHN;Tanz CRND; Charles H Tator, M.D, Principal Investigator — Toronto Western Hopsital,UHN
Locations (1):
- Canadian Concussion Centre, Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No